CLINICAL TRIAL: NCT00237666
Title: An Open-Label, Flexible-Dose Trial of the Safety and Efficacy of Geodon in Non-Rapid-Cycling Bipolar II Patients With Major Depression
Brief Title: Open-Label Study of Geodon in Non-Rapid Cycling Bipolar II Patients With Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Medical Research Network (Other)
Collaborators: Liebowitz, Michael R., M.D. (Individual); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-3945-A 01
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2013-06-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-05

CONDITIONS: Bipolar II Disorder; Major Depressive Episode
Keywords: Bipolar II Disorder; Major Depressive Episode
MeSH Terms: conditions — Bipolar Disorder | interventions — ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ziprasidone (Experimental): Ziprasidone monotherapy, 20-60 mg BID.
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Ziprasidone — Ziprasidone 20-60 mg BID, taken orally.
  Other Names: Geodon

SUMMARY:
The purpose of this study is to evaluate the antidepressant effectiveness of Geodon for the treatment of patients diagnosed with Bipolar II disorder who are currently experiencing a major depressive episode.

DETAILED DESCRIPTION:
Bipolar II disorder is largely unstudied, with much less known about its treatment in comparison to Bipolar I disorder. While established mood stabilizers treat and prevent subsequent episodes of hypomania, chronic or recurrent depressions are harder to treat or prevent. In general the treatment of depression in Bipolar II patients is often complicated and there is no clinical unanimity on what approaches to follow. Administration of proven antidepressants would seem most appropriate and are most often used, but their use often involves a number of difficulties. Among these are:

* antidepressant efficacy is established for unipolar patients and extrapolation to Bipolar II patients is done without empirical support
* Bipolar II patients can have switches into hypomanic behavior in response to antidepressant treatment given as monotherapy
* even when mood stabilizers are concomitantly given, switches to hypomanic states still occur when antidepressants are added
* antidepressants can cause cycle acceleration or induce rapid cycling when given to Bipolar II patients
* non-response and loss of response are common reactions to antidepressants in Bipolar II patients

This study will also assess the tolerability of Geodon in the treatment of patients diagnosed with Bipolar II disorder who currently meet criteria for a Major Depressive Episode by examining the incidence of adverse events and the withdrawal rate due to adverse events.

This will be an open-label study. Subjects will be treated for 8 weeks with Geodon, starting at a dose of 20 mg twice per day. The maximum dose will be 60 mg twice per day. Subjects will have a physical exam, electrocardiogram (ECG), standard laboratory tests and a urine drug screen at the screen visit.

Efficacy evaluations will include 17-item Hamilton Depression Scale, Hamilton Anxiety Scale (HAM-D), Montgomery-Asberg Depression Rating Scale, and the Young Mania Rating Scale. Social outcome will be measured with a quality-of-life scale (the Q-LES-Q). Overall efficacy will be rated using the Clinical Global Severity and Improvement Scales.

ELIGIBILITY:
Inclusion Criteria:

* patients will meet DSM-IV criteria for Bipolar II Disorder, with at least one hypomanic episode as documented in the medical history or provided by an informant, or have evidence of a clear diagnosis of hypomania
* patients will currently be experiencing a major depressive episode of 2 or more weeks, but less than 12 months duration
* minimum score of 18 on the 17-item HAM-D at screen and baseline

Exclusion Criteria:

* patients will not meet criteria for Bipolar I or Schizoaffective Disorder or Schizophrenia
* patients may have co-morbid anxiety or other Axis I disorders as long as depression dominates the clinical picture
* Suicidal ideation or history that makes participation in a clinical trial unduly risky
* unstable medical conditions or any abnormality in thyroid function
* patients with a QTc of 450msec or greater on the initial ECG
* patients requiring concomitant psychotropic drugs will not be eligible, although patients on such drugs who can undergo washout will be eligible. such patients must have discontinued psychoactive drugs at least 2 weeks before beginning study, with 4 weeks for fluoxetine and depot neuroleptics
* the use of Zolpidem 5-10 mg as needed will be permitted for patients suffering from insomnia, but cannot be taken the night before a scheduled assessment
* patients with dementia or substance abuse in the last 6 months
* pregnant or lactating women will be excluded, as will those not using adequate forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Liebowitz, MD, Principal Investigator — Medical Research Network, L.L.C.
Locations (2):
- United States (2):
  - Medical Research Network, L.L.C., New York, New York
  - The Mech Center, Plano, Texas

REFERENCES:
- See also: Study Site Information — http://www.medicalresearchnetwork.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at three research centers, located in: New York, NY; Plano, TX; and Seattle, WA. Subjects were recruited over a 37 month period.
Pre-assignment Details: The planned and actual study population was 30 patients, 18 years of age or older, who met DSM-IV criteria for bipolar II disorder with a history of at least one hypomanic episode.
Groups:
- Ziprasidone: Patients will receive 8 weeks of active treatment with ziprasidone, initiated at 20mg BID. Depending on tolerability and clinical response, the dosage can be titrated up to a maximum of 60mg BID per day. Dosage can be lowered or temporarily stopped if necessary because of adverse events.
Period: Overall Study
Arm/Group | Ziprasidone
Started | 30
Completed | 24
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.61 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is the Comparison of Baseline and Week 8 Endpoint in the 17-item HAM-D Total Scores
Description: Hamilton Depression Rating Scale, measuring depression symptoms; possible total scores ranging from 0-54, with higher scores indicating greater severity of symptoms.
Time Frame: Week 8
Population: Per protocol, the number of participants for analysis was 30 randomized subjects; data analyzed at Week 8 or Last Observation Carried Forward for the 6 subjects who dropped out before completion.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Ziprasidone: Ziprasidone 20-60 mg BID
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Scores on a scale
  Baseline HAM-D | 23.1 (3.49)
  Week 8 HAM-D | 10.57 (7.61)
Statistical Analysis 1: Comparison: Ziprasidone; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Mean Change From Baseline in the Hamilton Anxiety Scale (HAM-A)
Description: Hamilton Anxiety Rating Scale, measuring anxiety symptoms; possible total scores ranging from 0-30, with higher scores indicating greater severity of anxiety.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Scores on a scale
  Baseline HAM-A | 19.47 (4.10)
  Week 8 HAM-A | 10.69 (7.09)

3. Secondary Outcome: Mean Change From Baseline in the Montgomery-Asberg Depression Rating Scale
Description: Montgomery-Åsberg Depression Rating Scale, measuring depression symptoms; possible total scores ranging from 0-60, with higher scores indicating greater severity of depression.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Scores on a scale
  Baseline MADRS | 28.47 (4.96)
  Week 8 MADRS | 13.21 (8.99)

4. Secondary Outcome: Percentage of Subjects With Clinical Global Inventory (CGI) Global Improvement Score of 1 or 2
Description: Clinical Global Impression of Improvement scale: one item, measuring overall improvement of illness; possible scores range from 1-7, with lower scores representing greater improvement.
  18 subjects (60%) were responders (defined as having a CGI-I scores of 1 or 2 at Week 8/study endpoint) by the end of the trial.
Time Frame: Week 8
Measure: Number (95% Confidence Interval); unit: percentage of subjects with CGI-I </=2
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
percentage of subjects with CGI-I </=2 | 60 [42 to 77]

5. Secondary Outcome: Mean Change From Baseline in the CGI-Severity of Illness (CGI-S) Score at Study Endpoint
Description: Clinical Global Impression of Severity scale: one item, measuring overall severity of illness; possible scores range from 1-7, with higher scores representing greater severity of illness.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Score on a scale
  Baseline CGI-S | 4.27 (0.42)
  Week 8 CGI-S | 2.33 (1.13)

6. Secondary Outcome: Mean Change From Baseline in the Total Score of the Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q)
Description: Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) scale consists of 14 items; possible scores range from 14-70 with higher scores indicating greater quality of life and satisfaction.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Scores on a scale
  Baseline Q-LES-Q | 35.07 (7.34)
  Week 8 Q-LES-Q | 48.25 (12.97)

7. Secondary Outcome: Mean Change From Baseline in the Total Score of the Beck Depression Inventory (BDI)
Description: Beck Depression Inventory, self-rated scale measuring depression symptoms; possible total scores ranging from 0-63, with higher scores indicating greater severity of depression.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ziprasidone
Number analyzed (Participants) | 30
Scores on a scale
  Baseline BDI | 27.9 (9.78)
  Week 8 BDI | 15.0 (11.82)

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Ziprasidone
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ziprasidone (N=30)
White Blood Cell Count Decreased (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziprasidone (N=30)
Headache (General disorders) | 7
Drowsiness (General disorders) | 7
Insomnia (General disorders) | 6
Fatigue (General disorders) | 3
Gastrointestinal Upset (Gastrointestinal disorders) | 3
Dry Mouth (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No